CLINICAL TRIAL: NCT06839066
Title: A Phase II Study to Evaluate the Efficacy and Safety of HLX43 (Anti-PD-L1 ADC) in Subjects With Recurrent/Metastatic Nasopharyngeal Carcinoma (NPC) Failed or Intolerance to Second-line Therapy
Brief Title: A Phase II Study to Evaluate HLX43 in Subjects With Recurrent/Metastatic Nasopharyngeal Carcinoma Failed or Intolerance to Second-line Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX43-NPC201
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
Keywords: HLX43; Nasopharyngeal Carcinoma; anti-PD-L1 ADC
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HLX43 DOSE 1 (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), until disease progression and loss of benifit, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first).
  Interventions: Drug: HLX43 DOSE 1
- HLX43 DOSE 2 (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), until disease progression and loss of benifit, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first).
  Interventions: Drug: HLX43 DOSE 2
- HLX43 DOSE 3 (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), until disease progression and loss of benifit, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first).
  Interventions: Drug: HLX43 DOSE 3

INTERVENTIONS:
Drug: HLX43 DOSE 1 — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Arms: HLX43 DOSE 1
Drug: HLX43 DOSE 2 — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Arms: HLX43 DOSE 2
Drug: HLX43 DOSE 3 — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Arms: HLX43 DOSE 3

SUMMARY:
The study is to explore the reasonable dosage and to evaluate the efficacy, safety and tolerability of HLX43 (Anti-PD-L1 ADC) in patients with recurrent/metastatic Nasopharyngeal Carcinoma (NPC) who failed or are intolerant to second-line herapy.

DETAILED DESCRIPTION:
This study is an open-label phase II clinical study to explore the reasonable dosage and to evaluate the efficacy, safety and tolerability of HLX43 (Anti-PD-L1 ADC) in patients with recurrent/metastatic Nasopharyngeal Carcinoma (NPC) who failed or are intolerant to second-line therapy.

In this study, eligible subjects will be randomized at 1:1:1 ratio, and the patients will be administered with HLX43 at three different doses via intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the study content, procedures, and potential adverse reactions before the trial, sign the informed consent form (ICF), voluntarily participate in the trial, and be able to complete the study per the protocol requirements;
2. Age ≥ 18 years at the time of signing the ICF, regardless of gender;
3. Histologically or cytologically confirmed recurrent/metastatic nasopharyngeal carcinoma;
4. Recurrent/metastatic nasopharyngeal carcinoma patients who have failed or are intolerant to at least two prior lines of chemotherapy (including at least one platinum-based regimen) and PD-1/PD-L1 inhibitor therapy. Intolerance is defined as experiencing CTCAE ≥ grade 3 adverse events;
5. At least one measurable lesion per RECIST v1.1 within 4 weeks before randomization;
6. Willing to provide archived (preferably within 2 years) or fresh tumor tissue specimens for the detection of PD-L1 expression.
7. At least 4 weeks (or 5 half-lives, whichever is shorter) since last major surgery, medical device treatment, radiotherapy (except palliative bone radiotherapy), cytotoxic chemotherapy, immunotherapy, or biological therapy; ≥2 weeks since last hormonal therapy or small molecule targeted therapy; ≥1 week since last traditional Chinese medicine treatment with anti-tumor indications or minor surgery; with treatment-related adverse events recovered to CTCAE v5.0 ≤ grade 1 (except grade 2 peripheral neuropathy and alopecia);
8. ECOG performance status 0-1 within 1 week before randomization;
9. Expected survival ≥ 3 months；
10. Adequate organ function within 1 week before randomization (no blood transfusion or colony-stimulating factors within 14 days prior to first dose)
11. Fertile participants must use ≥1 highly effective contraceptive method during the trial and for ≥6 months after last dose; females of childbearing potential must have negative pregnancy test within 7 days before enrollment.

Exclusion Criteria:

1. Recurrent nasopharyngeal carcinoma candidates eligible for curative local therapy (surgery or radiotherapy).
2. Imaging showing tumor invasion/encasement of major thoracic/cervical/pharyngeal blood vessels (may be exempted if investigators confirm no impact on trial participation).
3. History of other malignancies within 2 years prior to randomization (except radically treated early-stage malignancies).
4. Previous ≥Grade 3 immune-related adverse events during immunotherapy.
5. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
6. Symptomatic/untreated/progressing CNS or leptomeningeal metastases.
7. History of ≥Grade 3 radiation pneumonitis; steroid-requiring (non-infectious) interstitial lung disease (ILD), current ILD, or ILD unexcludable by imaging; or severe respiratory impairment from pulmonary disease.
8. Poorly controlled cardiovascular/cerebrovascular conditions including.
9. Candidates for organ/marrow transplantation or previous transplant recipients.
10. Active systemic infections requiring IV antibiotics within 2 weeks pre-randomization.
11. Use of strong CYP2D6/CYP3A inhibitors/inducers within 2 weeks pre-randomization.
12. Systemic corticosteroid use (>10mg prednisone/day equivalent) or immunosuppressants within 2 weeks pre-randomization. Exceptions: Topical/ocular/intra-articular/nasal/inhaled steroids; short-term prophylactic use for contrast agents.
13. Active/suspected autoimmune diseases. Exceptions: Hypothyroid patients on thyroid replacement; controlled type 1 diabetes with insulin.
14. Live/attenuated vaccines within 4 weeks pre-randomization (inactivated influenza vaccines permitted).
15. History of severe hypersensitivity to biologics/monoclonal antibodies or trial drug components.
16. Active tuberculosis.
17. Immunodeficiency disorders (HIV-positive or congenital/acquired immune deficiencies).
18. Active HBV/HCV infection or co-infection:
19. Pregnant/lactating women.
20. Investigators' judgment of clinical/lab abnormalities or other factors making participation inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2026-11-22 (Estimated); Study Completion 2027-11-22 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 24 week
  Objective response rate (ORR) (assessed by INV per RECIST v1.1)
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Defined as the time (in months) from randomization to the first confirmed and documented progressive disease or death (whichever occurs first) as assessed by INV per RECIST v1.1.

SECONDARY OUTCOMES:
ORR | up to 24 week
  Objective response rate (ORR) (assessed by the IRRC per RECIST v1.1)
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Defined as the time (in months) from randomization to the first confirmed and documented progressive disease or death (whichever occurs first) as assessed by the IRRC per RECIST v1.1.
OS | From randomization to death from any cause (up to approximately 18 months)
  Overall Survival
Incidence and severity of adverse events (AEs) | time from the date of the first dose of study drug until 90 days after last dose, assessed up to 18 months
  severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version [v] 5.0

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Zhongshan City People's Hospital, Guangzhou, Guangdong
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen, Shenzhen, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Guizhou Medical University Cancer Hospital, Guiyang, Guizhou
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang